CLINICAL TRIAL: NCT06736470
Title: Surgical Suction Aspirates Fluorescence Measurement
Acronym: ATM GBM
Status: Recruiting | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: Marginum Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 5252665
Record Dates: First submitted 2024-11-20; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Gliomas; High-grade Glioma
Keywords: aspirate tissue monitoring; high-grade glioma; 5-ALA; fluorescence-guided surgery; neurosurgery
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 5-ALA: Patients who are prescribed 5-ALA (n=13)
- No 5-ALA: Patients who are not prescribed 5-ALA (n=7)

SUMMARY:
Gliomas are tumors that occur in all ages; they include the most common malign primary central nervous system tumors in developed countries. Gliomas are often aggressive, and their recommended treatment is surgical resection and chemoradiation. Complete tumor removal is challenging because of diffuse cell growth and the proximity of functionally critical tissues. Surgeons use 5-aminolevulinic acid (5-ALA) drug-induced fluorescence to visually detect tumor cells, which improves resection rates and delays tumor progression. Tumor cells are often left unnoticed because of visual obstacles or weak fluorescence, which may lead to local recurrence and reoperations. Surgical suction devices are used to remove cancerous tissues, but so far the suction aspirate tissues have not been routinely used in tissue detection. This single-center observational study compares experts' visual detection of 5-ALA-induced fluorescence and fluorescence detected from the surgical suction waste. The fluorescence from the suction waste will not be reported back to the surgeon.

DETAILED DESCRIPTION:
During glioma surgery, the diffuse boundary between healthy tissue and tumor is localized using 5-ALA drug-enhanced fluorescence of cancer cells. Visual fluorescence-based tissue recognition technique using 5-ALA has been shown to improve the rate of tumor removal and slow disease progression. To see the fluorescence typical of cancer, a special light source is needed in the operating microscope. In typical blue light, the fluorescence is visible, but it is more difficult detect anatomical landmarks, such as cerebral blood vessels and cranial nerves, which makes them vulnerable to injuries. Tumor cells can also be unnoticed because of visual obstacles or weak fluorescence, which may lead to local recurrence and reoperations. Unintended tumor remnants are frequent even though many other auxiliary techniques such as MRI guidance, neuronavigation, ultrasound and neurophysiological monitoring are used.

This single center observational study investigates a novel medical device's performance to detect 5-ALA (PpIX) fluorescence from the surgical suction waste. The fluorescence detected by the device is compared to expert's visual evaluation of fluorescence using an operating microscope. The comparison includes the device's feedback, operating videos under blue and white light, anatomical location and the results of histopathological analysis.

In total twenty-five (n=25) patients referred for resection surgery for suspected glioma or its recurrence at the Kuopio University Hospital. The patients are prescribed oral 5-ALA preoperatively according to the institution's practices and the suspected disease. Due to reasons not related to this study (lack of indication), some patients are not administered with 5-ALA. These patients are "control" patients providing reference data from brain tissues without exogenous fluorescent drugs to verify the device's safety and performance.

Informed written consent will be obtained from patients to participate in the study on the new surgical device. The clinical trial is approved by the local research ethics committees and approved by the Finnish Medicines Agency (Fimea). The investigated device is not CE-marked.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to neurosurgery department for surgical resection of a potential glioma
* Aged 18 years old or older
* Informed consent obtained

Exclusion Criteria:

* Patient belongs to the following vulnerable groups: children, pregnant, prisoners or intellectually disabled,,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Wellbeing Services County of North Savo region with a suspected glioma.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual fluorescence | 1 day (during surgical operation)
  Operating surgeon's evaluation of the presence of visual fluorescence in each scene. The expert panel's opinion of the presence of visual fluorescence in each scene of the operating video.
Fluorescence detected by the intestigational device | 1 day (during surgical operation)
  Fluorescence detected by the investigational device is compared against expert's visual detection.

CONTACTS AND LOCATIONS:
Overall Officials: Antti-Pekka Elomaa, Docent, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No
Potential GDPR limitations.